CLINICAL TRIAL: NCT07047807
Title: PDAC-PATHWAYS: A Digital Informational and Supportive Care App for Patients Initiating Neoadjuvant Therapy for Pancreatic Ductal Adenocarcinoma
Acronym: PDAC-PATHWAYS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kelsey S. Lau-Min, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-350
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: PDAC - Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDAC-PATHWAYS (Experimental): PDAC-PATHWAYS is an informational and supportive care app for patients initiating neoadjuvant therapy for PDAC.
  Interventions: Behavioral: PDAC-PATHWAYS
- Usual care (Active Comparator): Participants randomized to usual care will receive routine treatment with their oncology clinicians.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: PDAC-PATHWAYS — A digital app for patients initiating neoadjuvant therapy for PDAC
  Arms: PDAC-PATHWAYS
Other: Usual Care — Routine treatment
  Arms: Usual care

SUMMARY:
This study aims to refine and pilot test PDAC-PATHWAYS, a digital informational and supportive care app for patients who are initiating neoadjuvant therapy for pancreatic ductal adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
There are two parts of this study. Study Part 1 is an open pilot study to refine PDAC-PATHWAYS prior to larger-scale testing in a randomized controlled trial (RCT) setting. Study Part 1 is purely descriptive, as the investigators will use the data to refine PDAC-PATHWAYS before proceeding to Study Part 2.

Study Part 2 is a pilot RCT to assess the feasibility and acceptability of conducting a randomized trial of PDAC-PATHWAYS versus usual care. Participants will complete a baseline survey and then be randomized to PDAC-PATHWAYS versus usual care. This record reflects the clinical trial component (Study Part 2), as feasibility and acceptability outcomes will be collected for this phase only.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* Within 8 weeks of a documented decision to pursue neoadjuvant therapy for newly diagnosed, non-metastatic PDAC
* Able to comprehend and speak English

Exclusion Criteria:

* Comorbid health condition that would interfere with study participation, as identified by the cancer care team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Enrollment rate | 10 weeks
  ≥50% enrollment among consecutive eligible patients
Feasibility: intervention completion rate | 10 weeks
  ≥60% completion of at least three of the five app modules among those assigned to the intervention

SECONDARY OUTCOMES:
Acceptability | 10 weeks
  ≥75% of patients in the intervention arm reporting Client Satisfaction Questionnaire-8 scores above the midpoint score of 20 on a scale from 8-32 (higher scores indicate higher satisfaction)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General HospitaL, Boston, Massachusetts, United States